CLINICAL TRIAL: NCT00450060
Title: Postlumbar Puncture Complaints After Lumbar Punctures in Children and Adolescents: Frequency and Impact by Compariosn of Two Needle Designs
Brief Title: Juvenile Postlumbar Puncture Headache After Puncture With Needles With Quincke Tip or With Sprotte Tip
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PLPH-01/07
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2007-03

CONDITIONS: Headache
Keywords: postlumbar puncture headache; atraumatic needle; Sprotte; Quincke; lumbar puncture; headache; backache
MeSH Terms: conditions — Headache; Back Pain | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: lumbar puncture with Quincke-design needles
Device: lumbar puncture with Sprotte-design needles

SUMMARY:
The purpose of this study is to compare postlumbar puncture complaints as headache or backache after lumbar puncture with needles with Quincke design or with Sprotte design in children and adolescents.

DETAILED DESCRIPTION:
After lumbar puncture patients may develop complaints as position dependent headache, other headache or backache. Several though not all studies in adults showed that the frequency of complaints can be reduced by using non-traumatic Sprotte-design needles instead of cutting Quincke-design needles. In children and adolescents there are no comparable data published. In most pediatric hospitals in Germany Quincke needles are used.

Comparison: Children and adolescents from 4 to 18 years of age who have to undergo a lumbar puncture are randomly attributed to puncture with Quincke needle or with Sprotte needle. During the following days headache (main criterium), position-dependent headache, backache, vomitus, and malaise are noted. Pain is measured with a visual analogue scale/faces scale.

ELIGIBILITY:
Inclusion Criteria:

* lumbar puncture necessary for diagnostic reasons

Exclusion Criteria:

* intrathecal instillation at lumbar puncture
* patients in whom severity of disease make it impossible to judge endpoint criteria

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150
Dates: Start 2007-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
headache frequency
headache intensity

SECONDARY OUTCOMES:
position dependent-headache frequency
position dependent-headache intensity
backache frequency
backache intensity
practicability of needle designs (multiple punctures necessary?, longer lasting?

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Ebinger, DM, Study Chair — University Pediatric Hospital Heidelberg
Locations (2):
- Germany (2):
  - University Pediatric Hospital, Heidelberg
  - Klinik für Kinderheilkunde und Jugendmedizin, Heilbronn

REFERENCES:
- [Background] Ebinger F, Kosel C, Pietz J, Rating D. Headache and backache after lumbar puncture in children and adolescents: a prospective study. Pediatrics. 2004 Jun;113(6):1588-92. doi: 10.1542/peds.113.6.1588. PMID 15173478
- [Background] Ebinger F, Kosel C, Pietz J, Rating D. Strict bed rest following lumbar puncture in children and adolescents is of no benefit. Neurology. 2004 Mar 23;62(6):1003-5. doi: 10.1212/01.wnl.0000115387.67958.0f. PMID 15037713